CLINICAL TRIAL: NCT02636036
Title: A Phase I Multicenter, Open Label Study of Enadenotucirev Combined With PD-1 Inhibitor in Subjects With Metastatic or Advanced Epithelial Tumors
Brief Title: Phase I Study of Enadenotucirev and PD-1 Inhibitor in Subjects With Metastatic or Advanced Epithelial Tumors
Acronym: SPICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ColoAd1-1003
Record Dates: First submitted 2015-11-20; First posted 2015-12-21 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer; Squamous Cell Carcinoma of the Head and Neck; Epithelial Tumor
Keywords: metastatic; epithelial; advanced
MeSH Terms: conditions — Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma; Neoplasm Metastasis | interventions — enadenotucirev; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- enadenotucirev and nivolumab (Experimental)
  Interventions: Biological: enadenotucirev; Biological: nivolumab

INTERVENTIONS:
Biological: enadenotucirev
Biological: nivolumab

SUMMARY:
This is a Phase I multicenter, open label, nonrandomized study of enadenotucirev administered in combination with nivolumab in subjects with metastatic or advanced epithelial tumors (with focus on CRC, SCCHN, escalation phase), not responding to standard therapy.

DETAILED DESCRIPTION:
To characterise the safety and tolerability of enadenotucirev administered in combination with nivolumab in subjects with metastatic or advanced epithelial tumours.

A dose escalation phase is conducted in subjects with solid tumors of epithelial origin not responding to standard therapy to establish the MTD/MFD and optimum dosing schedule of the enadenotucirev and nivolumab combination treatment.

A dose expansion phase will further outline the dose level and schedule of enadenotucirev and nivolumab combination treatment and investigate signals of efficacy in three cohorts of subjects with specific epithelial tumour types.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females aged 18 years or over
* Disease status: - Diagnosis of metastatic or advanced CRC, UCC, SCCHN, salivary gland cancer or NSCLC not responding to standard therapy or for whom no standard treatment exists
* For patients who have received prior PD-1 / PD-L1 therapy (Cohorts 7A and 7B and dose expansion phase only): Prior PD-1 / PD-L1 inhibitor therapy in current line of treatment for ≥6 weeks and ≤4 months, with best response of stable disease or progressive disease
* ECOG performance status 0 or 1
* Predicted life expectancy of 3 months or more
* Ability to comply with study procedures in the Investigator's opinion
* Recovered to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies Adequate lung function
* Adequate renal function
* Adequate hepatic function
* Adequate bone marrow function
* Adequate coagulation tests: PT and aPTT within normal range or international normalized ratio (INR) ≤1.5
* Meeting reproductive status requirements
* Subjects must provide written informed consent to participate
* Willing to consent to tumour biopsies during the study

Exclusion Criteria:

* Pregnant or breastfeeding females
* Known history or evidence of significant immunodeficiency due to underlying illness
* Splenectomy
* Prior allogeneic or autologous bone marrow or organ transplantation
* Any history of renal disease, renal injury or auto-immune disease.
* History of idiopathic pulmonary fibrosis, drug induced pneumonitis, evidence of active pneumonia or pneumonitis on computed tomography scan
* Clinically or radiologically suspected, or evidence of, lymphangitic carcinomatosis
* Active infections requiring antibiotics, physician monitoring or recurrent fevers >100.4˚F (38.0˚C) associated with a clinical diagnosis of active infection
* Active viral disease or positive test for hepatitis B virus using hepatitis B surface antigen test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid or HCV antibody test indicating acute or chronic infection. Positive test for HIV or AIDS; testing is not required in the absence of history
* Use of the following antiviral agents: ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to the first dose of study treatment; or pegylated interferon in the 4 weeks before the first dose of study treatment
* For Cohort 1 to 6:Prior treatment with PD-1 and programmed death ligand (PD-L)1 inhibitors
* For Cohorts 7A and 7B and dose expansion phase: History of Grade >2 or currently uncontrolled immune-related AEs while being treated with PD-1 / PD-L1 inhibitors
* For Cohorts 7A and 7B and dose expansion phase: Patients with progressive disease with ≥50% increase in disease burden from start of PD-1 / PD-L1 inhibitor therapy in the most recent line of treatment are excluded
* Major surgery or treatment with any chemotherapy (bisphosphonate therapy or treatment with receptor activator of nuclear factor kappa-Β l(RANK)-ligand inhibitors for metastatic bone disease is permitted), biologics for cancer or investigational therapy in the 28 days before the first dose of study treatment (patients with prior cytotoxic or investigational products <3 weeks prior to study treatment might be eligible after discussion between the Investigator and Medical Monitor, if toxicities from the prior treatment have been resolved to NCI CTCAE Grade 1 and decision is supported by the half-life of previous therapy). All toxicities attributed to prior anti-cancer therapy other than alopecia must have resolved to Grade 1 or baseline before the first dose of study treatment. Patients with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll Note: This does not apply to anti-PD-1 / PD-L1 if in the patient's current line of therapy, and anti-PD-1 / PD-L1 treatment may continue during screening
* Other prior malignancy active within the previous 3 years except for local or organ confined early stage cancer that has been definitively treated with curative intent, does not require ongoing treatment, has no evidence of residual disease and has a negligible risk of recurrence and is therefore unlikely to interfere with the primary and secondary endpoints of the study, including response rate and safety
* Symptomatic brain metastases or any leptomeningeal metastasis that is symptomatic and/or requires treatment. Patients with brain metastases are eligible if these have been locally treated (surgery, radiotherapy). There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalent) for at least 14 days before the first dose of study treatment. Both surgery and or radiotherapy must have been completed at least 2 weeks before first dose of study treatment
* Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results
* Known allergy to enadenotucirev, nivolumab or their excipients
* Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
* Dependence on continuous supplemental oxygen use
* History of myocardial infarction or significant cardiovascular or cerebrovascular event in the 12 months before the first dose of study treatment
* An increased risk due to tumour flare, as assessed by the Investigator (e.g. an initial increase in tumour size that may lead to intestinal obstruction, obstruction of the ureter or airway)
* Penetrating tumour infiltration of major blood vessels, pericardium, gastrointestinal tract or other hollow organs that may lead to perforation due to tumour necrosis
* History of DVT or pulmonary embolus in the 12 months before the first dose of study treatment
* History of significant bleeding requiring hospitalization in the 12 months before the first dose of study treatment
* Patients receiving therapeutic or prophylactic anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events (safety and tolerability) in study of enadenotucirev administered in combination with a PD-1 inhibitor | 12 months
  Review of adverse events including serious adverse events (SAEs), adverse events meeting protocol defined DLT criteria, adverse events leading to study treatment or study discontinuation, and adverse events resulting in death
Maximum Tolerated and/or Maximum Feasible Dose | 12 months
  Maximum tolerated dose (MTD) / maximum feasible dose (MFD) of enadenotucirev administered IV in combination with nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lillie, MD, Study Director — Psioxus Theraputics
Locations (6):
- United States (6):
  - University of Arizona Cancer Center, 1515 North Campbell Ave., Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, 1500 E Duarte Str., Duarte, California
  - UCLA Medical Center, 10945 Le Conte Ave, Ste. 3360, Santa Monica, California
  - Horizon Oncology Research, 1345 Unity Place, Suite 365, Lafayette, Indiana
  - Henry Ford Hospital, 2799 West Grand Blvd., Detroit, Michigan
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fakih M, Harb W, Mahadevan D, Babiker H, Berlin J, Lillie T, Krige D, Carter J, Cox C, Patel M, Parfitt L, Powell M, Rosen L. Safety and efficacy of the tumor-selective adenovirus enadenotucirev, in combination with nivolumab, in patients with advanced/metastatic epithelial cancer: a phase I clinical trial (SPICE). J Immunother Cancer. 2023 Apr;11(4):e006561. doi: 10.1136/jitc-2022-006561. PMID 37094988
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458